CLINICAL TRIAL: NCT00996541
Title: Diverting Homeless Youth From Chronic Homelessness and Risk for HIV
Brief Title: Support To Reunite Involve and Value Each Other
Acronym: STRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01MH070322-05 (NIH); 5R01MH070322-05 (NIH)
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Family Relations; Runaway Behavior; Risky Sexual Behavior; Substance Use
Keywords: Runaway youth; Homeless youth; Family intervention; Family functioning; HIV risk behavior; HIV Seronegativity
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: STRIVE family intervention
- Control (Placebo Comparator)
  Interventions: Behavioral: STRIVE family intervention

INTERVENTIONS:
Behavioral: STRIVE family intervention — Adolescent and parent attend a 5-session family-oriented cognitive-behavioral intervention aimed at giving runaway youths and their parents the tools to effectively deal with conflict.

SUMMARY:
Runaway and homeless youth are at risk for HIV based upon their rates of substance use, particularly injection drug use, unprotected sexual intercourse, multiple partners, and sexually transmitted diseases. Risk increases as the time away from home increases. STRIVE is a family intervention aimed at increasing residential stability, decreasing runaway episodes, and decreasing HIV risk. Families are randomly assigned to a cognitive-behavioral skills-building intervention consisting of five weekly sessions delivered at family homes, or are assigned to standard care. Sessions are aimed at increasing problem solving, role clarity, and positive interactions. It is hypothesized that the intervention will result in improved family dynamics, less runaway behavior, and less risky behavior.

ELIGIBILITY:
Inclusion Criteria:

* Youth: Age 12-17 who ran away or were told to leave home within the past 6 months. Must provide assent and parent/guardian must provide informed consent.
* Parent/guardian: must be parent/guardian of participating youth who ran away. Must provide informed consent.

Exclusion Criteria:

* Youth: total time away from home exceeds 12 months. Obvious cognitive impairment. Sexual or physical abuse from the parent/guardian. Lack of assent/consent.
* Parent/guardian: obvious cognitive impairment. Lack of consent.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Improved residential stability | Assessed up to 24 months

SECONDARY OUTCOMES:
Reduced HIV risk behavior | Up to 24 months

REFERENCES:
- [Result] Milburn NG, Iribarren FJ, Rice E, Lightfoot M, Solorio R, Rotheram-Borus MJ, Desmond K, Lee A, Alexander K, Maresca K, Eastmen K, Arnold EM, Duan N. A family intervention to reduce sexual risk behavior, substance use, and delinquency among newly homeless youth. J Adolesc Health. 2012 Apr;50(4):358-64. doi: 10.1016/j.jadohealth.2011.08.009. Epub 2011 Oct 26. PMID 22443839